CLINICAL TRIAL: NCT00530439
Title: Lifestyle and Pregnancy: The Clinical Effect of Lifestyle Intervention During Pregnancy in Obese Women
Acronym: LiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Christina Vinter, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 029
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-04

CONDITIONS: Maternal Obesity; Gestational Weight Gain; Obstetric Complications
MeSH Terms: conditions — Pregnancy in Obesity; Gestational Weight Gain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): physical activity, dietetic counselling
  Interventions: Other: Lifestyle intervention; Behavioral: Physical activity, dietetic counselling
- Control (No Intervention)
  Interventions: Other: Control

INTERVENTIONS:
Other: Lifestyle intervention — Dietician counselling and physical training
  Arms: Lifestyle intervention
Other: Control — Repeated measuring of maternal weight gain, blood samples and ultrasound
  Arms: Control
Behavioral: Physical activity, dietetic counselling — The active intervention consisted of two major components: dietary counseling and physical activity. Dietary counseling was performed by trained dieticians on four separate occasions at 15, 20, 28 and 35 weeks gestation.
  Energy requirements for each participant were individually estimated according to weight and level of activity during pregnancy. Women in the active intervention group were encouraged to be moderately physically active 30-60 minutes a day.Women in this group also had free full time membership in a fitness center for six months. In the fitness centers they had closed training classes with trained physiotherapists for one hour each week.
  Arms: Lifestyle intervention

SUMMARY:
Obesity is a serious and increasing health problem in the Western World with about one third of all pregnant women in Denmark being overweight. Among these are more than 11% severe obese.

Obesity in pregnancy is related to higher maternal morbidity and perinatal morbidity and mortality. Observational studies indicate that the rate of pregnancy complications among obese pregnant women can be limited if weight gain during pregnancy is restricted.

Aims of the trial is to study the effects of diet and physical training during pregnancy among Danish obese women. Also to describe the metabolic effects of lifestyle intervention during pregnancy.

360 obese pregnant women with Body Mass Index (BMI) > 30 are randomized to lifestyle intervention group or control group. The intervention is composed of individual dietician counselling and physical training. The physical training includes weekly aerobic exercises in a fitness center and lifestyle coaching in small groups.

Both groups will be examined during pregnancy with extra ultrasound scanning of the fetus, blood pressure, and metabolic markers. All women receive vitamin supplementation to assure sufficient intake.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant
* BMI >/= 30 and </= 45

Exclusion Criteria:

* Chronic diseases
* Not Danish speaking
* Abuse of alcohol or drugs
* Preterm delivery in earlier pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A. Vinter, Ph.d. Student, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Vinter CA, Tanvig MH, Christensen MH, Ovesen PG, Jorgensen JS, Andersen MS, McIntyre HD, Jensen DM. Lifestyle Intervention in Danish Obese Pregnant Women With Early Gestational Diabetes Mellitus According to WHO 2013 Criteria Does Not Change Pregnancy Outcomes: Results From the LiP (Lifestyle in Pregnancy) Study. Diabetes Care. 2018 Oct;41(10):2079-2085. doi: 10.2337/dc18-0808. Epub 2018 Jul 30. PMID 30061318
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Beck-Nielsen H, Christesen HT, Jensen DM. Effects of lifestyle intervention in pregnancy and anthropometrics at birth on offspring metabolic profile at 2.8 years: results from the Lifestyle in Pregnancy and Offspring (LiPO) study. J Clin Endocrinol Metab. 2015 Jan;100(1):175-83. doi: 10.1210/jc.2014-2675. PMID 25343235
- [Derived] Vinter CA, Jorgensen JS, Ovesen P, Beck-Nielsen H, Skytthe A, Jensen DM. Metabolic effects of lifestyle intervention in obese pregnant women. Results from the randomized controlled trial 'Lifestyle in Pregnancy' (LiP). Diabet Med. 2014 Nov;31(11):1323-30. doi: 10.1111/dme.12548. Epub 2014 Jul 23. PMID 24989831
- [Derived] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Tanvig M, Lamont RF, Jorgensen JS. Postpartum weight retention and breastfeeding among obese women from the randomized controlled Lifestyle in Pregnancy (LiP) trial. Acta Obstet Gynecol Scand. 2014 Aug;93(8):794-801. doi: 10.1111/aogs.12429. Epub 2014 Jun 13. PMID 24834792
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Lamont RF, Beck-Nielsen H, Christesen HT, Jensen DM. Anthropometrics and body composition by dual energy X-ray in children of obese women: a follow-up of a randomized controlled trial (the Lifestyle in Pregnancy and Offspring [LiPO] study). PLoS One. 2014 Feb 24;9(2):e89590. doi: 10.1371/journal.pone.0089590. eCollection 2014. PMID 24586896
- [Derived] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Intervention | Control
Started | 180 | 180
Completed | 150 | 154
Not Completed | 30 | 26
Not completed — GDM | 9 | 3
Not completed — Withdraw | 18 | 14
Not completed — Missed abortion | 1 | 4
Not completed — Misclassification | 2 | 0
Not completed — Twin pregnancy | 0 | 2
Not completed — Severe malformation/abortion | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Control | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 180 | 360
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.6 (4.35) | 29.05 (4.12) | 29.3 (4.2)
Age Continuous [Median (Inter-Quartile Range); unit: Years] | 29 [27 to 32] | 29 [26 to 32] | 29 [26 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 180 | 360
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 180 | 180 | 360

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Section
Time Frame: At delivery
Reporting Status: Not Posted

2. Primary Outcome: Preeclampsia/Pregnancy Induced Hypertension
Time Frame: Delivery
Reporting Status: Not Posted

3. Primary Outcome: Gestational Diabetes Mellitus
Time Frame: Delivery
Reporting Status: Not Posted

4. Primary Outcome: Large for Gestational Age
Time Frame: Delivery
Reporting Status: Not Posted

5. Primary Outcome: Neonatal Intensive Care Unit
Time Frame: Within 1 month postpartum
Reporting Status: Not Posted

6. Secondary Outcome: Metabolic Markers
Time Frame: Until 6 months post partum
Reporting Status: Not Posted

7. Primary Outcome: Gestational Weight Gain
Description: Weight at gestational week 35 - weight by inclusion
Time Frame: Gestational week 35
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Lifestyle Intervention | Control
Number analyzed (Participants) | 144 | 148
kg | 7.0 [4.7 to 10.6] | 8.6 [5.7 to 11.5]
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Control; Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Lifestyle Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No